CLINICAL TRIAL: NCT07281521
Title: Safety & Effectiveness of the CardioWave Pulsed Field Ablation System With the QuickShot Nav Large-Area Focal Catheter for Ablation of Persistent Atrial Fibrillation
Brief Title: Ablation With the PFA System With a Large-Area Focal Catheter for the Treatment of Persistent Atrial Fibrillation
Acronym: Quick AF
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: CardioFocus (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 25-6647
Record Dates: First submitted 2025-12-04; First posted 2025-12-15 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Persistant Atrial Fibrillation
Keywords: ablation; pulsed field ablation; atrial fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- Pulsed Field Ablation Treatment (Experimental): The treatment arm will undergo catheter ablation for persistent atrial fibrillation with the PFA system with a Large-Area Focal Catheter
  Interventions: Device: pulsed field ablation

INTERVENTIONS:
Device: pulsed field ablation — pulsed field ablation with a large-area focal catheter

SUMMARY:
The study evaluates the safety and effectiveness of the investigational QuickShot Nav configuration of the CardioWave System for focal catheter ablation of persistent atrial fibrillation (PerAF).

DETAILED DESCRIPTION:
This is a prospective, single-arm, multi-center, clinical study. The study will be conducted at up to 4 centers in Europe. Up to 200 participants will be enrolled and treated.

Participants enrolled in Phase A and Phase B will be exited from the study upon completion of the remapping procedure hospital discharge. Participants enrolled in Phase C will be followed through 12 months. All eligible patients who provide written informed consent will be treated with the study device.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of recurrent symptomatic paroxysmal AF (PAF) or persistent AF (PerAF) with the following documentation:

   Paroxysmal AF (Phase A participants)
   1. Physician's note indicating symptoms consistent with recurrent symptomatic PAF AND
   2. At least one documented episode of AF captured continuously on 12-lead ECG, or for at least 30 seconds on transtelephonic monitor (TTM), Holter monitor, telemetry strip, or similar within 12 months prior to enrollment

   Persistent AF (Phase A, B, and C participants)
   1. Physician's note indicating symptoms consistent with recurrent symptomatic PerAF AND
   2. Any 24-hour ECG recording of continuous AF within 12 months prior to enrollment OR
   3. Two ECGs from any form of rhythm monitoring showing continuous AF taken at least 7 days apart within 12 months prior to enrollment OR
   4. History of ≥2 direct current cardioversion (DCCV) performed within 12 months prior to enrollment
2. Failure or intolerance of at least one antiarrhythmic drug (AAD) (Class I - IV) for AF, as evidenced by recurrent symptomatic PerAF or intolerable side effects due to the AAD
3. Age 18 through 75 years-old on the day of enrollment
4. Patient is indicated for an ablation procedure according to society guidelines or study site practice
5. Patient is willing and able to give informed consent and is willing, able, and committed to participate in baseline and follow-up evaluations for the full duration of the study

Exclusion Criteria:

1. Long-standing persistent AF (continuous AF sustained > 1 year)
2. AF secondary to electrolyte imbalance, thyroid disease, alcohol abuse, or other reversible/non-cardiac causes
3. Prior cardiac ablation or surgical procedure (including left atrial appendage (LAA) device or occlusion, or valvular cardiac procedure)
4. Planned LAA closure procedure or implant of a permanent pacemaker, biventricular pacemaker, or any type of implantable cardiac defibrillator (with or without biventricular pacing function) for any time during study participation
5. Presence of any permanent pacemaker, biventricular pacemaker, or implantable cardiac defibrillator (with or without biventricular pacing function) that cannot be programmed, per the manufacturer's recommendations, during the ablation procedure
6. Patient cannot be removed from AADs for reasons other than AF, which includes participants with Wolff-Parkinson-White (WPW) Syndrome and participants with a history of ventricular tachycardia (VT)
7. Presence of any IVC filters
8. Presence of an interatrial baffle or patch
9. Presence of any pulmonary vein stents
10. Pre-existing pulmonary vein stenosis
11. Pre-existing hemidiaphragmatic paralysis
12. Atrial or ventricular septal defect closure
13. Atrial myxoma
14. Presence of any mechanical or biologic prosthetic heart valve
15. Hemodynamically significant valvular disease as determined by the Investigator
16. History of pericarditis
17. History of Rheumatic heart disease
18. History of thromboembolic event within 6 months prior to Index Ablation Procedure or evidence of intracardiac thrombus at time of the Index Ablation Procedure
19. Any of the following events within 3 months prior to the Index Ablation Procedure:

    * Myocardial infarction
    * Unstable angina
    * Percutaneous coronary intervention
    * Heart surgery including coronary artery bypass grafting
    * Heart failure hospitalization
    * Cerebral ischemic event (stroke or transient ischemic attack (TIA))
    * Clinically significant bleeding requiring surgical intervention
    * Pericardial effusion
    * Ventriculotomy or atriotomy
20. New York Heart Association (NYHA) Class IV congestive heart failure
21. Documented left ventricular ejection fraction (LVEF) ≤35% measured by acceptable cardiac testing (e.g., TTE, cardiac CT, etc.) within 6 months prior to enrollment
22. Hypertrophic cardiomyopathy
23. Primary pulmonary hypertension
24. Significant or symptomatic hypotension
25. Thrombocytosis, thrombocytopenia
26. Contraindication to, or unwillingness to use, systemic anticoagulation
27. Patient contraindicated for CT or MRI
28. Sensitivity to contrast media not controlled by premedication
29. Women known to be pregnant or breastfeeding, or any women of childbearing potential who are not on a reliable form of birth regulation method or abstinence
30. Patient is participating in any other potentially confounding research
31. Serious or untreated medical conditions that would prevent participation in the study, interfere with assessment or therapy, or confound data or is interpretation, including but not limited to:

    * Solid organ or hematologic transplant, or currently being evaluated for organ transplant
    * Severe lung disease, pulmonary hypertension, or any lung disease involving abnormal blood gases or significant dyspnea
    * Chronic renal insufficiency with eGFR <50 mL/min/1.73 m2, any history of renal dialysis, or history of renal transplant
    * Active malignancy or history of treated cancer within 24 months prior to enrollment
    * History of severe esophageal ulcers, strictures, esophagitis, esophageal structural abnormality, and uncontrolled/untreated gastroesophageal reflux disease (GERD)
    * Active systemic infection
    * Clinically significant psychological condition that, in the Investigator's opinion, would prohibit the participant's ability to meet the protocol requirements
    * Predicted life expectancy <1 year

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-02-27 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Primary Safety Endpoint - Rate of Primary Serious Adverse Events | 7 days (unless otherwise specified)
  The rate of participants with at least 1 of the following Primary Serious Adverse Events occurring within 7 days unless otherwise specified:
  * Atrio-esophageal fistula (assessed at ≥60 days)
  * Cardiac perforation, tamponade, or pericardial effusion
  * Cerebrovascular accident (CVA)/stroke
  * Complete heart block
  * Death
  * Major vascular access complications/bleeding requiring surgical intervention or blood transfusion
  * Myocardial infarction
  * Pericarditis
  * Phrenic nerve injury resulting in persistent diaphragmatic paralysis (assessed at ≥60 days)
  * Pulmonary vein stenosis (assessed at ≥60 days)
  * Thromboembolism
  * Transient ischemic attack (TIA)
  * Vagal nerve injury/gastroparesis
Primary Effectiveness Endpoint - Acute Procedure Success | During procedure
  Percentage of treated pulmonary veins with documented PVI at the end of the index procedure using the study device only. Acute PVI will be assessed by the confirmation of entrance and/or exit block.
  • Inability to isolate a targeted pulmonary vein with the study device and requiring use of a non-study ablation device to complete PVI will count as an acute procedure failure.

SECONDARY OUTCOMES:
Chronic PVI Durability | 60 days post-procedure
  Percentage of treated pulmonary veins with documented PVI at the remapping procedure. Chronic PVI will be assessed by the confirmation of entrance and/or exit block for all pulmonary veins treated at the index procedure.
Acute Success of Additional Atrial Lesion Sets | During procedure
  Percentage of additional atrial lesion sets (PWI, CTI, mitral isthmus) with documented acute procedural success using the study device only.
12-Month Freedom from Atrial Arrhythmia | 12 months post-procedure
  Freedom from documented atrial arrhythmia (AF/AFL/AT) episodes ≥30 seconds duration, after the 60-day Blanking Period following the index ablation procedure, documented by trans-telephonic monitoring (TTM) or Holter monitor through 12 months follow-up.

CONTACTS AND LOCATIONS:
Locations (3):
- KBC Split, Split, Croatia
- Czechia (2):
  - St. Anne's University Hospital, Brno
  - Homolka, Prague

IPD SHARING:
Plan to Share IPD: No